CLINICAL TRIAL: NCT04858100
Title: Comparison Between Surgical Excision and "Wait and See" Approach in the Treatment of Oral Leukoplakia: a Randomized, Controlled Clinical Trial
Brief Title: Oral Potentially Malignant Disorders: Comparison Between Surgical Treatment and Wait and See Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giovanni Lodi, Associate Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LEUKO2020
Record Dates: First submitted 2021-03-02; First posted 2021-04-26 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Leukoplakia, Oral
Keywords: Oral Potentially Malignant Disorder; Oral carcinoma; Oral medicine; Cancer prevention
MeSH Terms: conditions — Leukoplakia, Oral; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Experimental): Each patient will receive the surgical excision of the lesion and subsequent follow-up
  Interventions: Procedure: Surgical excision of the lesion
- Wait and see (Active Comparator): Each patient will receive clinical follow-up of the lesion with periodical incisional tissue biopsy.
  Interventions: Other: Wait and see approach

INTERVENTIONS:
Procedure: Surgical excision of the lesion — The surgical removal of the lesion, performed within 3 months from the final diagnosis, will follow these steps:
  * local anesthesia
  * excision of the lesion with surgical blade or laser, according to the clinical case, paying attention to having at least 2 mm-free margins
  * silk or resorbable suture for wound closure
  The patient will be recall after 14 days for assessing the wound healing and after 30 days for providing and explaining him the histopahtological exam.
  The patient will receive a 3-6 month follow-up according to the clinical and histopathological case.
  Arms: Surgery
Other: Wait and see approach — The patient will receive a 3-6 month follow-up according to the clinical and histopathological case, with periodical incisional biopsy every 4 control visit.
  In case of OSCC onset during the first 3 months after the final diagnosis, the patient will be excluded since the oral cancer occurence will be considered as a misdiagnosis, more than a "true" malignat progression.
  Arms: Wait and see

SUMMARY:
This research protocol is comparing the effectiveness of surgical excision to the "wait and see" approach for the management of oral leukoplakia and erythroleukoplakia in prevention of oral squamous cell carcinoma onset.

DETAILED DESCRIPTION:
Different treatments have been proposed for the management of oral leukoplakia (OL) in order to prevent oral squamous cell carcinoma onset. However, there is still no consensus on the most effective approach for the patients affected by such oral potentially malignant disorders. Surgery is often performed, but there is no randomized clinical trial which demonstrates its real effectiveness in preventing oral cancer onset.

A recent RCT compared surgical treatment with "wait and see approach" care in patients with nondysplastic OL, assuming that regular clinical follow-up could be considered a reliable standard of care among patients with nondysplastic oral leukoplakias.

The purpose of this study is to evaluate effectiveness of surgical excision in treating OL and or reducing the onset of potential oral squamous cell carcinoma, with a follow-up of 5 years. This study will be the first RCT comparing the effectiveness of surgery to "wait and see approach" in the management of both dysplastic and nondysplastic oral leukoplakias.

ELIGIBILITY:
Inclusion Criteria:

* OL diagnosis should be confirmed by incisional diagnostic biopsy and subsequent histopathological analysis
* Subjects' age: 18 years or older
* Lesions' size: 3 cm maximum longitudinal size of the single lesion
* Lesions's location: oral areas with no surgical risk of damages to important anatomical structures such as nerves, salivary ducts and/or arteries.
* Ability to understand and to sign a written informed consent document

Exclusion Criteria:

* Previous oral cancer
* Head and neck radiotherapy
* Subjects under the age of 18
* Subjects affected by PVL (proliferative verrucous leukoplakia)
* High-risk of surgical damages to anatomical structures such as nerves, salivary ducts and/or arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Oral cancer incidence | every 3 or 6 months (according to the clinical case) up to 5 years
  Number of patients who will develop oral squamous cell carcinoma

SECONDARY OUTCOMES:
Time to malignant transformation from diagnosis | every 3 or 6 months (according to clinical case) up to 5 years
  Period of time required to develop malignancy
Quality of life after surgical excision | month 1 and month 6
  To evaluate the quality of life of patients affected by leukoplakia and treated with surgical excision, via Functional Intraoral Glasgow Scale (FIGS) questionnaire. FIGS is a simple point scale used to assess a patient's ability to speak, chew and swallow. Each of these functions is scored independently on a scale of 1-5, five being no disability and one meaning the patient has an inability to speak, chew, or swallow.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Lodi, PhD, DMD, Principal Investigator — University of Milan
Locations (2):
- Italy (2):
  - Università degli Studi di Torino Dental School, Turin, TO
  - University of Milan, Milan